CLINICAL TRIAL: NCT03137706
Title: Characterization of Mechanical Tissue Properties in Pancreas, Liver and Colon
Brief Title: Characterization of Mechanical Tissue Properties in Patients With Pancreatic, Liver, or Colon Cancer
Status: Terminated | Type: Observational
Why Stopped: Insufficient accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0S-16-1; NCI-2016-01955 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-16-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-04-29; First posted 2017-05-03 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Colon Carcinoma; Liver and Intrahepatic Bile Duct Carcinoma; Pancreatic Carcinoma
MeSH Terms: conditions — Colonic Neoplasms; Carcinoma, Hepatocellular; Pancreatic Neoplasms | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-correlative (tissue stiffness analysis): Patients undergo fresh tumor tissue collection at the time of surgery. The fresh tumor tissue samples are analyzed for tissue stiffness measurements using optical polarimeter device and cell viability using automated cell counter.
  Interventions: Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis; Other: Laboratory Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo fresh tumor tissue collection
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Laboratory Procedure — Tissue stiffness and cell viability analysis
  Other Names: Lab Test; Lab Tests; Laboratory Test; Test; Tests

SUMMARY:
This pilot research trial studies characterization of mechanical tissue properties in patients with pancreatic, liver, or colon cancer. Mechanical properties and stiffness of the cancerous tissue may be correlated with the standard pathology report that describes the stage of the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if our optical polarimeter device is able to measure tissue stiffness across several human cancer types ex vivo.

SECONDARY OBJECTIVES:

I. To describe the inter- and intra-tumor heterogeneity of tissue stiffness. II. To determine if the measurements made by the optical polarimeter device are non-destructive.

TERTIARY OBJECTIVES:

I. Perform multi-variable cross-correlation statistical analysis to determine relationships between: tissue stiffness characteristics, molecular level signatures, and cellular level properties, and if numbers permit, response to treatment.

OUTLINE:

Patients undergo fresh tumor tissue collection at the time of surgery. The fresh tumor tissue samples are analyzed for tissue stiffness measurements using an optical polarimeter device and cell viability using an automated cell counter.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgery to remove primary tumors in the pancreas, liver or colon and have not undergone any prior treatment
* Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Pregnant women will not be consented
* Patients that are unable to consent for surgery
* Primary liver tumors with cirrhosis will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgery to remove primary tumors in the pancreas, liver, or colon
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Young's modulus (stiffness) on fresh tissue | Up to 15 months
  A portable optical fiber polarimetric sensor device to measure the Young's modulus in tissue samples will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Mumenthaler, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided